CLINICAL TRIAL: NCT02045914
Title: Effect of Calcium Ionophore Solution on Fertilization Rate During ICSI Cycles of Poor Ovarian Reserve Patients
Brief Title: Calcium Ionophore Solution Can Increase Fertilization Rate in Patients During Intracytoplasmic Sperm Injection(ICSI) Who Have Poor Ovarian Reserve?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Pinar Caglar Aytac, Effect of calcium ionophore solution on fertilization rate during ICSI cycles of poor ovarian reserve patients, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KA1-191
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Fertilization Failure
Keywords: calcium ionophore; fertilization rate; poor ovarian reserve
MeSH Terms: interventions — Ionomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): the patients who have no intervention with calcium ionophore during ICSI cycle
- calcium ionophore (Experimental): the patients whose oocytes are incubated with calcium ionophore solution during ICSI cycle
  Interventions: Other: calcium ionophore solution

INTERVENTIONS:
Other: calcium ionophore solution — After microinjection of sperm into the oocyte, oocytes are incubated for 15 minutes in a 30 microlitre droplet of calcium ionomycin solution
  Other Names: GM 508 Cult-Active (Gynemed); ionomycin
  Arms: calcium ionophore

SUMMARY:
The aim of this study is to evaluate calcium ionophore solution on fertilization rate of patients during intracytoplasmic sperm injection who have poor ovarian reserve

DETAILED DESCRIPTION:
During ICSI cycle , female patients who have poor ovarian reserve have low oocyte numbers. So by calcium ionophore solution which we know that it can increase fertilization rate in males who have azospermia or globozoospermia. we planned to check if this solution can increase fertilization rate also in poor ovarian reserve patients?

ELIGIBILITY:
Inclusion Criteria:

* infertile couples who have no male factor infertility
* infertile females who are poor ovarian reserve

Exclusion Criteria:

* infertile couples who have male factor infertility
* infertile female who have endometriosis

Ages: 23 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
calcium ionophore solution effect on fertilization rate | 18 hours
  Before Intracytoplasmic sperm injection adding calcium ionophore solution to the medium can increase fertilization rate of oocytes or not?

SECONDARY OUTCOMES:
Calcium ionophore solution increase on going pregnancy rate | up to 21 weeks
  İf the calcium ionophore can increase fertilization rate , pregnancy rate up to 20 weeks, can increase or not?

OTHER OUTCOMES:
calcium ionophore can decrease fertilization rate | 18 hours
  To detect if calcium ionophore can affect fertilization rate in a reverse manner than expected

CONTACTS AND LOCATIONS:
Overall Officials: esra bulgan kilicdag, prof md, Study Director — Baskent University; Huriye Ayse Parlakgumus, md, Study Chair — Baskent University; Pinar Caglar Aytac, md, Principal Investigator — Baskent University; Cok Tayfun, md, Study Chair — Baskent University; Bulent Haydardedeoglu, assoc Prof, Study Chair — Baskent University; Erhan Simsek, md, Study Chair — Baskent University
Locations (1):
- baskent university obstetric and gynecology, reproductive endocrinology and IVF unit, Adana, Kisla, Turkey (Türkiye)

REFERENCES:
- [Derived] Caglar Aytac P, Kilicdag EB, Haydardedeoglu B, Simsek E, Cok T, Parlakgumus HA. Can calcium ionophore "use" in patients with diminished ovarian reserve increase fertilization and pregnancy rates? A randomized, controlled study. Fertil Steril. 2015 Nov;104(5):1168-74. doi: 10.1016/j.fertnstert.2015.07.1163. Epub 2015 Sep 3. PMID 26342247